CLINICAL TRIAL: NCT06252103
Title: Lactoferrin With Ferrous Gluconate Versus Ferrous Gluconate in Treatment of Iron Deficiency Anemia During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS298/2023
Record Dates: First submitted 2024-01-22; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-05

CONDITIONS: Lactoferrin With Ferrous Gluconate More Superior Than Ferrous Gluconate Alone in Treatment of Iron Deficiency Anemia
Keywords: iron deficiency anemia during pregnancy; ferrous gluconate; lactoferrin
MeSH Terms: interventions — ferrous gluconate; Lactoferrin

STUDY DESIGN:
Intervention Model Description: Total 40 females from 14 to 35 weeks of pregnancy with Hemoglobin level between 8.5 to 10.5 gm/dl, recruited from the obstetric inpatient/outpatient clinic at Ain Shams University, Maternity hospital.
  This study included two groups:
  Group I: 20 patients were given ferrous gluconate 300 mg (Ferrous-Gluconate®, tab.300mg glucofer, Egypt) two times daily.
  Group II: 20 patients were given lactoferrin 100mg (Pravotin-sachets®,100mg, Hygint, Egypt) with ferrous gluconate twice daily.
  hematological parameters (rise in hemoglobin) and the adverse effects of both drugs were studied at registration and after 4 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Active Comparator): the first group 20 patients will receive one tab of ferrous gluconate 300mg administered orally twice per day for 4 weeks (Ferrous-Gluconate®, tab.300mg glucofer, Egypt) two times daily.
  Interventions: Drug: Ferrous Gluconate 300 MG
- group II (Active Comparator): 20 patients were given lactoferrin 100mg (Pravotin-sachets®,100mg, Hygint, Egypt) with ferrous gluconate twice daily for 4 weeks Patients were assigned to take the medication orally; once daily before breakfast, and Pravotin (100 sachets were be dissolved each in ¼ glass of water and taken before breakfast). Patients were advised to avoid the intake of tea, coffee, milk, milk products, antacids and calcium preparation within 2 hours before or after iron capsules.
  Interventions: Drug: ferrous gluconate with lactoferrin

INTERVENTIONS:
Drug: Ferrous Gluconate 300 MG — iron salt one tab 300 mg contain 35 mg of elemental iron given 2 doses 600 mg per day
  Other Names: (Ferrous-Gluconate®, tab.300mg glucofer, Egypt
  Arms: group I
Drug: ferrous gluconate with lactoferrin — Lactoferrin is a glycoprotein from the transferrin family consist of 691 amino acids,Lactoferrin is a protein found in cow milk and human milk
  Other Names: Pravotin-sachets®,100mg, Hygint, Egypt) with ferrous gluconate twice daily.
  Arms: group II

SUMMARY:
Study Procedures:

All patients will undergo the following:

Informed consent will be obtained from all the participants in this study before enrolling in this study and all participants will be subjected to a detailed clinical assessment including: a detailed history, general, abdominal examinations, Investigations.

1. History taking:

   * Personal history: name, age, occupation and address.
   * Menstrual and obstetric history: Date of LMP, expected date of delivery which will be calculated according to Naegle's rule and gestational age. In addition to history of presence of any menstrual irregularities, duration.
   * Past History: of Anemia in previous pregnancy, other diseases like Thalassemia, sickle cell anemia, liver or renal diseases or any other condition that may affect hemoglobin.
2. Medical examination:

   * General: Assessment of complexion and vital data (blood pressure, pulse, capillary refill)
   * Abdominal examination to assess fundal height.
3. Investigations to perform will include:

Laboratory: Complete blood count (microcytic hypochromic anemia) Imaging: Ultrasound to assess biometry to exclude fetal growth restriction. Women will be divided in two groups with 20 in each group, the first group will receive one tab of ferrous gluconate 300mg administered orally twice per day for 4 weeks and the second group will receive lactoferrin sachets 100mg with ferrous gluconate 300mg twice per day for 4 weeks Patients were assigned to take the medication orally; once daily before breakfast, and Pravotin (100 sachets were be dissolved each in ¼ glass of water and taken before breakfast). Patients were advised to avoid the intake of tea, coffee, milk, milk products, antacids and calcium preparation within 2 hours before or after iron capsules.

Women will be told to record side effects as nausea, vomiting, abdominal discomfort and constipation.

Women will have a blood sample (CBC) withdrawn after 2 to 4 weeks to assess rise in pregnant anemia.

DETAILED DESCRIPTION:
This study included two groups:

Group I: 20 patients were given ferrous gluconate 300 mg (Ferrous-Gluconate®, tab.300mg glucofer, Egypt) two times daily.

Group II: 20 patients were given lactoferrin 100mg (Pravotin-sachets®,100mg, Hygint, Egypt) with ferrous gluconate twice daily.

hematological parameters (rise in hemoglobin) and the adverse effects of both drugs were studied at registration and after 4 weeks

ELIGIBILITY:
* The study will include women with the following inclusion and exclusion criteria:

Inclusion criteria:

1. Pregnant women with single fetus
2. Microcytic hypochromic anemia, mild anemia Hb 10 to 10.5 g/dl) and moderate anemia (Hb 7 to 9.9 g/dl)
3. Gestational age (14 - 35 weeks)
4. Serum ferritin level <24 ng/dl

Exclusion Criteria:

1. Associated chronic medical disorder (CKD, liver disease, peptic ulcer and chronic blood loss).
2. Associated bleeding disorder
3. Anaemia requiring blood tranfusion (Hb < 7gm/dL)
4. Hypersensitivity to iron preparations
5. Haemoglobinopathies (G6PD, thalassemias, sickle cell disease)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
• Hemoglobin (Hb) level | 4 weeks
  hemoglobin will be measured before and after treatment by 4 weeks (HB in gm/dl)
serum ferritin | 4 weeks
  serum ferritin will be measured before and after treatment by 4 weeks (ferritin in ug/l )

SECONDARY OUTCOMES:
gastrointestinal side effects | 4 weeks
  (nausea , vomiting , constipation ) will be assessed before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: AMR Saad, doctoral, Study Director — faculty of medicine Ain shams university
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt